CLINICAL TRIAL: NCT00582023
Title: CHAI Study: Coping, HIV, and Affect Interview Study
Brief Title: Role of Positive Affect in Adjustment to HIV
Acronym: CHAI
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: CHAI 971423990; R01MH068170 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
Keywords: HIV; coping; emotion; affect; HIV infection; Complimentary therapies
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine the role of emotion and mood in the context of HIV.

DETAILED DESCRIPTION:
A growing body of literature indicates that positive affect may have a unique adaptive role in the process of adjustment to chronic stress, independent of the effects of negative affects like depression. The overarching goal of this research is to provide evidence and direction for the development of interventions for people with HIV that include a focus on positive affect. To this end, this study will document the occurrence, predictors, and consequences of positive affect during the 18 months post-notification of HIV+ serostatus.

ELIGIBILITY:
Inclusion Criteria:

* Have been informed they were HIV positive within the past two months
* Speak English
* Be 18 years or older
* Have the ability to provide informed consent to be a research participant

Exclusion Criteria:

* Severe cognitive impairment
* Active psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults newly diagnosed with HIV in the San Franicsco Bay Area.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2004-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Well being | 18 month follow-up
Physical & Mental Health | 18 months
Coping Response | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Judith Moskowitz, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Osher Center for Integrative Medicine, UCSF, San Francisco, California, United States